CLINICAL TRIAL: NCT05189340
Title: Development of Discharge Education Video for Solid Organ Transplant Recipients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00303596
Record Dates: First submitted 2021-12-29; First posted 2022-01-12 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Educational Activities; Organ Transplants

STUDY DESIGN:
Intervention Model Description: Patients in the standard of care arm will be enrolled through a specified date (currently targeting late February 2022, at which time enrolled patients will be included in the intervention group until data collection ceases in late April
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patients in the Standard of Care arm will receive pharmacist discharge education via fully in-person education as is currently being done.
- Intervention (Experimental): Patients in the Intervention arm will have access to pre-recorded educational videos covering key educational points. Patients will also have in-person interaction with pharmacists to address additional questions not covered in the videos.
  Interventions: Other: Educational Videos

INTERVENTIONS:
Other: Educational Videos — Series of six videos each covering a specific aspect of post-transplant care related to medication use or monitoring
  Arms: Intervention

SUMMARY:
Audiovisual teaching aids can play a significant role for the retention of new material and help overcome barriers such as the physical presence or time restrictions of an instructor. In a clinical setting, multimedia health education can offer an advantage over traditional didactic teaching by engaging patients through visual content and unlimited accessibility.

A critical factor to long-term survival of solid organ transplant recipients is compliance to post-transplantation medication and follow-up patient care. Transplant pharmacists serve on multidisciplinary care teams as the medication experts that provide discharge education to recipients and caregivers often at the bedside. The adoption of digital multimedia content for patient education can increase engagement of diverse learning styles while simultaneously reducing potential time conflicts in hospital practice. This study contributes to the literature by assessing the effectiveness of discharge education video(s) on patient satisfaction and knowledge levels which are currently limited.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are solid organ transplant recipients at Johns Hopkins Hospital
* Patients who are being managed by an adult solid-organ transplant surgical service
* Patients who can speak and read the English language

Exclusion Criteria:

* Patients with language access services needs will be excluded
* Patients who do not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-04-11 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Patient Transplant Medication and Care Knowledge | Pre- and post-education; pre-education assessment will be completed as soon as feasible after transplant (estimate 1-3 days) and consent; post-education assessment will be completed as soon as is feasible after initial education (estimate 0-2 days)
  Change in performance pre and post-education based on responses to questionnaire
Patient Satisfaction with Educational Method | As soon as feasible post-education, in concert with post-education knowledge assessment (estimate 0-2 days)
  Difference in satisfaction as determined by response to questionnaire post education. A single question score from 1 to 10 will be used, with 10 being highest satisfaction and 1 being the lowest level of satisfaction

SECONDARY OUTCOMES:
Pharmacist Time Requirement | As soon as feasible post-education (estimate 0-2 days)
  Time required by pharmacist for education

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Whisler, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No